CLINICAL TRIAL: NCT05685017
Title: Adiponectin, ICAM-1, VCAM-1 Levels and Metabolic Syndrome in Obese Adolescents
Acronym: ICAM; VCAM
Status: Completed | Type: Observational
Sponsor: Universitas Airlangga (Other)
Responsible Party: Principal Investigator, Andy Darma, MD, Principal Investigator on Gastroenterology, Universitas Airlangga
Other Study IDs: Secondary ID
Record Dates: First submitted 2023-01-01; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Obesity; Abdominal Obesity; Metabolic Syndrome; Hypertension; Hypertriglyceridemia; HDL Cholesterol, Low Serum; Hyperglycemia
MeSH Terms: conditions — Obesity; Obesity, Abdominal; Metabolic Syndrome; Hypertension; Hypertriglyceridemia; Hypoalphalipoproteinemias; Hyperglycemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Blood samples were withdrawn via vena cubitus as much as 5 ml by the trained analyst, and placed on vacutainer with EDTA. After that, the vacutainer was replaced in icebox to transport to the laboratory. Blood analysis including: lipid profile, fasting blood glucose, fasting insulin and adiponectin using the ELISA method in the laboratory. Intercellular Adhesion Molecule-1 (ICAM-1) was analyzed using Human intercellular adhesion molecule 1 Elisa kit (Bioassay Technology Laboratory). while sVCAM-1 was analysed using Human vascular cell adhesion molecule-1 Elisa kit (Bioassay Technology Laboratory).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metablic syndrome vs. non-metabolic syndrome: Obese adolescents were grouped on MetS vs. non-MetS based on The International Diabetic Federation criteria
  Interventions: Diagnostic Test: Nur Aisiyah Widjaja

INTERVENTIONS:
Diagnostic Test: Nur Aisiyah Widjaja — Blood analysis for ICAM-1, VCAM-1, blood fasting insulin, lipid profile, fasting blood glucose and adiponectin investigation
  Other Names: Suhasta Nova; Leonardo Alexander Caesar

SUMMARY:
Adipose tissue secreting a number of adipokines which regulate insulin sensitivity, energy metabolism and vascular homeostasis, so the dysfunction of adipose tissue is linked with the incidence of obesity accompanied with insulin resistance, hypertension and cardiovascular disease (1). Obesity is known to alters the expression of adipokines due to the adipose tissue hypertrophy (2), including adiponectin, in which able to exert a potent anti-inflammatory and vascular protective effect (2).

It has been proposed that adiponectin acts to prevent the vascular dysfunction due to obesity and diabetes by improves insulin sensitivity and metabolic profiles to reduce the risk factors for cardiovascular disease and protects the vasculature through its pleiotropic actions on endothelial cells, endothelial progenitor cells, smooth muscle cells and macrophages (1). The concentrations of adiponectin of 5 to 25 mg/mL had a significant inhibitory effect on the expression of monocyte adhesion and adhesion molecule induced by TNF-α in vitro. Atherosclerosis is an inflammatory disease in which adhesion molecules on arterial endothelial cells are responsible for the accumulation of monocytes/macrophages and T lymphocytes. While obesity is low-grade inflammation in which make a contribution on endothelial dysfunction by increasing the oxygen-derived free radicals (ROS) due to adipocyte hypertrophy, leads to an endoplasmic reticulum (ER) stress and mitochondrial dysfunction (3). Adiponectin is accumulated in the vasculature, and it reduced on obesity due to suppression by TNF-α and lead to adiponectin-deficiency which stimulate the significant increases of Vascular cell adhesion protein 1 (VCAM-1) and Intercellular Adhesion Molecule 1 (ICAM-1) or known as CD54 in aortic intima (4).

Here we investigate the level of adiponectin, ICAM-1, VCAM-1 with the incidence of MetS in obese adolescents.

DETAILED DESCRIPTION:
A cross sectional study with healthy obese adolescents aged 13 until 18 years old were conducted during October 2019 to January 2020. Obesity was determined based on body mass index (BMI) for age based on gender > percentile 95th of CDC growth chart 2000.

Body weight was measured using Seca Robusta 813 digital scale in standing position, by stepping on the scale. While Body height was measured using Seca 206 Body Meter. Height was measured from the vertex of the head to the heel in standing position. Waist circumference and hip circumference were measured using Seca 201 measuring tape. Waist circumference was measured by wrapping the measuring tape around the subject's stomach, at the midpoint between the lowest rib and the endpoint of the iliac crest upon expiration, in line with the navel. Hip circumference was measured by asking the subjects to keep the feet together, then wrapping the measuring tape around the widest part of hips, at the point of the greatest gluteal protuberance. The subjects were measured using light cloth without food wear and other accessories such as belt, hat, or hair accessories, etc.

Blood pressure was measure using Omron Automatic Blood Pressure Monitor HEM-8712 (Omron Health Care Co., Ltd, Japan) by placing the cuff on the right arm, then pull and tighten it according to the size if the arm. After it was installed correctly (fasten and did not move), the power button on the digital tension tool was pressed, and then the microprocessor started to drive air pressure into the cuff, and then the value of blood pressures will appear in the manometer tube column.

Metabolic syndrome criteria were determined using The International Diabetic Federation criteria18:

1. For adolescent aged 10-16 years old: if there was a central obesity (waist circumference > 90th percentile based on WHO waist circumference table. For boys at the circumference of > 88 cm, and ≥ 85 cm for girls) accompanied with at least 2 other signs below:

   * Blood pressure > 90th percentile (systole ≥130/diastole ≥ 85 mmHg).
   * Hypertriglyceridemia, if the triglyceride levels > 110 mg/dl.
   * Low level HDL-c, if the HDL-c levels < 40 mg/dl, and < 50 mg/dl for girls.
   * Hyperglycaemia, if fasting blood glucose (FBG) levels was > 110 mg/dl.
2. For adolescent aged more than 16 years old: if there was a central obesity (waist circumference > 90th percentile based on WHO waist circumference table. For boys at the circumference of > 94 cm, and ≥ 80 cm for girls) accompanied with at least 2 other signs below:

   * Blood pressure > 90th percentile (systole ≥130/diastole ≥ 85 mmHg).
   * Hypertriglyceridemia, if the triglyceride levels ≥ 150 mg/dl.
   * Low level HDL-c, if the HDL-c levels <40 mg/dl for boys, and < 50 mg/dl for girls.
   * Hyperglycaemia, if fasting blood glucose (FBG) levels was ≥ 100 mg/dl19. Blood samples were withdrawn via vena cubitus as much as 5 ml by the trained analysts, and placed on vacutainer with EDTA. After that, the vacutainer was replaced in icebox to transport to the laboratory. Blood analysis include: lipid profile, fasting blood glucose, fasting insulin and adiponectin using the ELISA method in the laboratory. Intercellular Adhesion Molecule-1 (ICAM-1) was analyzed using Human intercellular adhesion molecule 1 Elisa kit (Bioassay Technology Laboratory). while sVCAM-1 was analysed using Human vascular cell adhesion molecule-1 Elisa kit (Bioassay Technology Laboratory).

Statistical analysis conducted were test of normality and homogeneity test, Anova/ Kruskal-Wallis, Independent sample T-test/Mann-Whitney U test, and Spearman correlation, and determined as significant if p value<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Obesity
* Healthy (no medication treatment)

Exclusion Criteria:

* Taking corticosteroids or dyslipidemia medication
* Smoking or drinking (consuming alcohol)
* Taking antibiotics or hormonal therapy
* Autoimmune disease
* Endocrinology disorders

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The subjects were obese adolescents who were studied at Junior and Senior High School in Surabaya and Sidoarjo, East Java, Indonesia
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
ICAM-1 levels | 4 months
  Intercellular Adhesion Molecule 1 also known as CD54 was measured Human intercellular adhesion molecule 1 Elisa kit (Bioassay Technology Laboratory), stated as pg/ml (mean +/- SD)
VCAM-1 | 4 months
  Vascular cell adhesion molecule 1 was measured using Human vascular cell adhesion molecule-1 Elisa kit (Bioassay Technology Laboratory), stated as pg/ml (mean +/- SD)
Adiponectin | 4 months
  For Adiponectin, ICAM-1 and VCAM-1 analysis, the blood that has been taken was not immediately analysed. The blood was centrifuged to remove the serum, and then stored at -70°C until the analysis was performed in the laboratory. Adiponectin was analysed using using Human Adiponectin Elisa kit (Bioassay Technology Laboratory), stated as ng/ml (mean +/- SD)

SECONDARY OUTCOMES:
Physical Measurements: Body weight | 4 months
  body weight was measured using Seca Robusta 813 digital scale in standing position by stepping on the scale. The subjects were asked to use light clothes without footwear or accessories. Stated as kg (mean +/- SD)
Physical Measurements: Body height | 4 months
  Body height was measured using Seca 206 Body Meter. Height was measured from the vertex of the head to the heel in standing position without footwear or accessories such as hat

OTHER OUTCOMES:
Physical Measurements: Waist Circumference | 4 months
  Waist circumference was measured by wrapping the measuring tape (Seca 201 measuring tape),around the subject's stomach, at the midpoint between the lowest rib and the endpoint of the iliac crest upon expiration, in line with the navel. Stated as cm (mean +/- SD)
Physical Measurements: Hip Circumference | 4 months
  Hip circumference was measured by asking the subjects to keep the feet together, then wrapping the measuring tape (Seca 201 measuring tape) around the widest part of hips, at the point of the greatest gluteal protuberance, stated as cm (mean +/- SD)
Blood Pressure: Systole and diastole | 4 months
  Blood pressure was measured using Omron Automatic Blood Pressure Monitor HEM-8712, Omron Health Care Co., Ltd, Japan. The cuff was placed on the right arm, then pull and tighten it according to the size if the arm. After it was installed correctly (fasten and did not move), the power button on the digital tension tool was pressed, and then the microprocessor started to drive air pressure into the cuff, and then the value of blood pressures will appear in the manometer tube column. Stated as mmHg (mean +/- SD)
Blood biochemistry: HDL-c levels | 4 months
  The HDL-c levels were analysed by a designated medical laboratory after withdrawn, stated as mg/dl (mean +/- SD)
Blood biochemistry: Triglyceride levels | 4 months
  The triglyceride levels were analysed by a designated medical laboratory after withdrawn, stated as mg/dl (mean +/- SD)
Blood biochemistry: Fasting blood glucose levels | 4 months
  Fasting blood glucose levels were analysed by a designated medical laboratory after withdrawn, stated as mg/dl (mean +/- SD)
Blood biochemistry: Fasting insulin levels | 4 months
  Fasting insulin levels were analysed by a designated medical laboratory after withdrawn, stated as mg/dl (mean +/- SD)

CONTACTS AND LOCATIONS:
Overall Officials: Andy Darma, Paediatrician, Principal Investigator — Child Health Departement Airlangga University
Locations (1):
- Institute of Tropical Disease (ITD) Airlangga University, Campus C, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No